CLINICAL TRIAL: NCT04624568
Title: Papilocare®: Effects on Regression of Histologically Confirmed Cervical Intraepithelial Lesions 1 and Tolerance.
Acronym: PAPILOCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRO-2020-13
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Squamous Intraepithelial Lesions of the Cervix; Human Papilloma Virus Infection; Cervix Lesion
Keywords: Cervical lesion; Cervical intraepithelial lesions 1; CIN1; Low grade lesion; Colposcopy; Cervical cytology; Human Papillomavirus; HPV infection; HPV testing; Vaginal gel; Papilocare®
MeSH Terms: conditions — Squamous Intraepithelial Lesions of the Cervix; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: clinical trial with 2 parallel groups :
  1. Treatment arm : Use of the vaginal gel for the first 6 months, then absence of treatment for the next 6 months until follow-up.
     * First month : 1 cannula of Papilocare® per day except the last 7 days of the month.
     * The next five months : alternate days except the last 7 days of the month.
  2. Control arm - Absence of treatment for 12 months.
  Inclusion of 150 patients, balanced randomization meaning 75 patients in each arm.
  Follow-up after 6 months : a cervical cytology and a HPV testing for each patient + listing how many patients suffer from vaginal discomfort for 6 months.
  Follow-up after 12 months : a cervical cytology and a HPV testing for each patient.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Papilocare group (Experimental): Papilocare® for 6 months according to the following schedule:
  1 self-applying single dose per day for 21 days over 28 during the first month, then 1 day over 2 during the following 5 months, with a 7-day break during the menstrual period. (This break must be respected even in menopausal women or women undergoing artificial amenorrhea (amenorrhea induced by certain contraceptives: implant, hormonal IUD, micro-progestogen).
  Interventions: Device: PAPILOCARE
- Control group (No Intervention): No treatment for 12 months. Smear and HPV test will be perform by all patients at 6 and 12 months

INTERVENTIONS:
Device: PAPILOCARE — Papilocare® is a self-administered vaginal gel. Its single-dose cannula contains hyaluronic acid and pre-biotics (Coriolus Versicolor) that would improve the re-epithelialization of the uterin cervix. By creating a protective film on the cervix, this gel could induce a favorable environment for regression of the cervical intraepithelial lesions 1 and for clearance of Human Papillomavirus.
  The specific approach related to our study would be to apply Papilocare® vaginal gel for 6 months for the treated group.
  Smear and HPV test will be perform by all patients at 6 and 12 months.
  Arms: Papilocare group

SUMMARY:
clinical trial comparing the regression rate after 12 months of histologically confirmed cervical intraepithelial lesions 1 in 2 parallel groups. One group using the vaginal gel Papilocare® for 6 months and one group without any treatment.

DETAILED DESCRIPTION:
Cervical cancer affects 3000 women and causes 1100 deaths every year in France. This type of cancer usually takes about 10 to 15 years to develop and has distinct precursor stages. Persistent infection by Human Papillomavirus is necessary for the development of these lesions.

Currently, when a colposcopy biopsy reveals low grade lesion, it is recommanded to make a new cervical cytology or HPV testing, 12 months later. No treatment is recommended over this period. However 11% of these lesions evolve from low to high grade.

Papilocare® is a vaginal gel that would improve the re-epithelialization of the uterine cervix. Creating a protective film on the cervix, it could induce a favorable environment for regression of the cervical intraepithelial lesions 1 and for clearance of Human Papillomavirus.

The goal of our study is to include 150 women with a histologically confirmed cervical intraepithelial lesions 1. Half of them will be using the vaginal gel Papilocare® for 6 month while the other half will not receive any treatment (as suggested by current recommendations). Each patient will have a cervical cytology and a HPV testing after 6 months and after 12 months. Therefore we will be able to compare the percentage of normalization of cervical cytology and HPV clearance for each group after 6 months and after 12 months.

Patients will visit the Orleans hospital once for the inclusion and twice for follow-ups after 6 months and 12 months.

If the use of Papilocare® really induces a significant regression of low grade lesions, this vaginal gel could be offered as soon as these lesions are histologically identified in order to stop its progress to high grade.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 years old or older.
* With histologically-confirmed cervical intraepithelial lesion 1 only, proven by colposcopy biopsy, done in the most suspiscious area.
* With complete colposcopy, performed less than 3 months prior the inclusion
* With confirmed ASC-US or LSIL cervical-cytology, performed less than 6 months prior the colposcopy.

Exclusion Criteria:

* Women under guardianship or curatorship
* Women under the protection of justice
* Women not affiliated with a social security system
* Pregnant woman (as vaginal gel has not been evaluated in pregnant women) Urinary dosing of BHCG will be performed on the day of inclusion for all women under 55 years of age and effective contraception is recommended during the study for all non-menopausal women.
* Immunodepressed women (HIV, immunosuppressive treatments ...)
* Woman using vaginal contraceptives (ring, spermicides, cervical cap; because of risk of interaction) NB: Papilocare is compatible with the use of condoms and intrauterine devices.
* Known allergy to one of the components
* Patients with low-grade histology with HSIL - ASC-H - AGC smear will not be included. The cyto-colposcopic discordance suggests a high-grade lesion that would not have been biopsied at colposcopy.
* Patients undergoing laser or conization treatment according to the recommendations of INCa 2016 will not be included; namely: persistence of CIN 1 for more than 24 months on at least 2 different colposcopies; high-grade squamous intraepithelial histological lesions; adenocarcinoma in situ.
* Participation in another interventional study

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-05-17 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
Cervical cytology normalization after 12 months. | Month 12
  Compare the normalization rate of the cervical cytology in each arm after 12 months.
  The difference will be considered statistically significant if the treatment group has a normalization rate of 25% or higher.
  An "unsatisfactory" smear in its realization will have to be repeated within 45 days.

SECONDARY OUTCOMES:
Cervical cytology normalization after 6 months. | Month 6
  Compare the normalization rate of the cervical cytology in each arm after 6 months.
HPV clearance after 6 months | Month 6
  2) Compare in each arm the rate of transition from a positive HPV testing at inclusion to a negative HPV testing after 6 months.
  The difference will be considered statistically significant if the treatment group has a clearance rate of 25% or higher.
HPV clearance after 12 months | Month 12
  2) Compare in each arm the rate of transition from a positive HPV testing at inclusion to a negative HPV testing after 12 months.
  The difference will be considered statistically significant if the treatment group has a clearance rate of 25% or higher.
Evaluation of tolerance of Papilocare vaginal gel | Month 6
  Compare in each group the number of episodes of vaginal discomfort over the first 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Helene GBAGUIDI, Dr, Principal Investigator — CHR ORLEANS
Locations (1):
- Centre Hospitalier Régional d'Orléans, France, Orléans, France

REFERENCES:
- [Background] Bosch FX, Lorincz A, Munoz N, Meijer CJ, Shah KV. The causal relation between human papillomavirus and cervical cancer. J Clin Pathol. 2002 Apr;55(4):244-65. doi: 10.1136/jcp.55.4.244. PMID 11919208
- [Background] Ostor AG. Natural history of cervical intraepithelial neoplasia: a critical review. Int J Gynecol Pathol. 1993 Apr;12(2):186-92. PMID 8463044
- [Background] Lousuebsakul V, Knutsen SM, Gram IT, Akin MR. Clinical impact of atypical squamous cells of undetermined significance. A cytohistologic comparison. Acta Cytol. 2000 Jan-Feb;44(1):23-30. doi: 10.1159/000326220. PMID 10667155
- [Result] Bansal N, Wright JD, Cohen CJ, Herzog TJ. Natural history of established low grade cervical intraepithelial (CIN 1) lesions. Anticancer Res. 2008 May-Jun;28(3B):1763-6. PMID 18630456